CLINICAL TRIAL: NCT03453164
Title: Combination of Checkpoint Inhibitor and Radiotherapy for Recurrent Gastric Cancer After Initial Treatment With Standard Therapy (CIRCUIT).
Brief Title: Checkpoint Inhibitor and Radiotherapy for Recurrent Gastric Cancer (CIRCUIT)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fukushima Medical University (Other)
Responsible Party: Principal Investigator, Koji Kono, Professor, Fukushima Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RK29040
Record Dates: First submitted 2018-02-21; First posted 2018-03-05 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Gastric Cancer
Keywords: Radiotherapy; anti-PD-1 antibody
MeSH Terms: conditions — Stomach Neoplasms | interventions — Radiotherapy; Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy + Nivolumab (Experimental): Localized short-term radiotherapy (22.5 Gy/5 fractions/5 days, Day 1-5) + nivolumab (starting on Day 15-22, a dose of 3 mg/kg (body weight) or 240 mg/body, every 2 weeks to a total of 6 courses)
  Interventions: Radiation: Radiotherapy; Drug: Nivolumab

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy of 22.5 Gy/5 fractions/5 days was given to a symptomatic lesion or the largest asymptomatic lesion suitable for irradiation from Day 1.
Drug: Nivolumab — Nivolumab was administered intravenously starting on Day 15-22 at a dose of 3 mg/kg (body weight) or 240 mg/body every 2 weeks to a total of 6 courses of administration.
  Other Names: Opdivo

SUMMARY:
This study aims to evaluate safety and efficacy of nivolumab (anti-PD-1 antibody), which is approved as tertiary therapy, and neoadjuvant short-term limited local radiotherapy in patients with unresectable recurrent gastric cancer who progressed (intolerance or PD) after standard treatment (primary and secondary chemotherapy) and have more than one lesion assessable in diagnostic imaging (one lesion must be >=2cm).

DETAILED DESCRIPTION:
In patients with unresectable recurrent gastric cancer who progressed (intolerance or PD) after standard treatment (primary and secondary chemotherapy) and have more than one lesion assessable in diagnostic imaging (one lesion must be >=2cm), localized short-term radiotherapy of 22.5 Gy/5 fractions/5 days is applied to a symptomatic lesion or the largest asymptomatic lesion suitable for irradiation (Day 1-5). Nivolumab is administered starting from Day 15-22 at a dose of 3 mg/kg (body wait) or 240 mg/body every 2 weeks to a total of 6 courses (end of intervention).

The patients are observed up to Day 180±14 and evaluated on Day 180±14 (end of study).

ELIGIBILITY:
Inclusion Criteria:

1. Unresectable advance or recurrent GC with intolerance or progression after standard treatment (primary and secondary chemotherapy).
2. More than one measurable lesion defined by RECIST guideline version 1.1 in diagnostic imaging (whole-body contrast-enhanced CT or PET-CT) within 14 days before entry, with at least one lesion >=2 cm.
3. Age: 20 =<
4. ECOG performance status (PS): 0-2
5. No contraindication for nivolumab (anti-PD-1 antibody) administration.
6. No contraindication for radiotherapy.
7. The most recent laboratory results within 14 days before study entry fulfill the following: WBC ≥3000/μl, neutrophil ≥1500/μl, hemoglobin ≥9.0g/dl, platelets ≥100,000/μl, total bilirubin ≤2.0 times the institutional standard upper limit (ISUL), AST (GOT) and ALT (GPT) ≤3.0 times ISUL (in case with liver metastasis, ≤5.0 times ISUL), serum creatinine ≤1.5 times ISUL or creatinine clearance ≥ 60 ml/min calculated with cockcroft-Gault equation.
8. Expected survival >=3 months.
9. Written informed consent is obtained from the patient prior to study enrollment.

Exclusion Criteria:

1. No tumor lesions that can be irradiated.
2. Metachronous and simultaneous overlapping cancers (excluding intraepithelial cancer of the uterine cervix, fully treated basal cell carcinoma of the skin, and malignant tumors that were treated more than 5 years ago and have not recurred).
3. A history of severe hypersensitivity reactions to other Ab products.
4. Taking immunosuppressive drugs or corticosteroids (prednisone or prednisolone equivalent ≥ 15 mg/day).
5. Active autoimmune diseases or a history of recurrent autoimmune diseases (patients with type-1 diabetes, hypothyroid controllable by hormone replacement therapy, and dermatosis without the need for systemic therapy are eligible).
6. Complications or history of interstitial pneumonia or pulmonary fibrosis diagnosed by imaging studies or clinical findings.
7. Presence of severe disease or medical conditions: severe nutritional deficiencies, transient ischemic attack within 180 days prior to enrollment, cerebral vascular attack within 180 days prior to enrollment, thrombus or thromboembolism within 180 days prior to enrollment, congestive heart failure (NYHA class III or IV), unstable angina, myocardial infarction within 12 months, severe arrhythmias requiring medication, conduction abnormalities such as AV block beyond the second degree, uncontrollable hypertension, liver cirrhosis (Child Class B or higher), mental disorders that may interfere with compliance with this study protocol, unstable diabetes, uncontrolled pericardial fluid, uncontrolled ascites, uncontrolled pleural effusions, diseases requiring anticoagulation therapy (excluding antiplatelet therapy including low-dose aspirin), and systemic infection with treatment.
8. Pregnant or lactating female.
9. Fertile female who are unwilling to use contraception.
10. Fertile male who are not willing to use contraception during study drug administration and for 7 months after study completion (if the partners are fertile females).
11. Prohibited previous treatment: within 56 days of registration; radioactive drugs (except radiopharmaceuticals for examination or diagnostic purposes), within 28 days of registration; corticosteroids (excluding temporary use and predonine or prednisolone equivalent ≤15 mg/day), immunosuppressant drugs, anti-cancer drugs, adhesive treatment of pleura or pericardium, surgery with general anesthesia, and unapproved drugs, within 14 days of registration; surgery with local or superficial anesthesia.
12. Participating in other clinical trials or clinical studies (excludes those without intervention).
13. A positive HIV antigen/Ab test or HTLV-1 Ab test.
14. History of treatment using ONO-4538, anti-PD-1 Ab, anti-PD-L1 Ab, anti-PD-L2 Ab, anti-CD137 Ab, anti-CTLA-4 Ab, or other Ab or drug therapies for T-cell regulation.
15. Determined by the investigator to be ineligible for participation in this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Koji Kono, Professor, Principal Investigator — Fukushima Medical University Hospital
Locations (1):
- Fukushima Medical University Hospital, Fukushima, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suzuki Y, Mimura K, Yoshimoto Y, Watanabe M, Ohkubo Y, Izawa S, Murata K, Fujii H, Nakano T, Kono K. Immunogenic tumor cell death induced by chemoradiotherapy in patients with esophageal squamous cell carcinoma. Cancer Res. 2012 Aug 15;72(16):3967-76. doi: 10.1158/0008-5472.CAN-12-0851. Epub 2012 Jun 14. PMID 22700877
- [Background] Yoshimoto Y, Suzuki Y, Mimura K, Ando K, Oike T, Sato H, Okonogi N, Maruyama T, Izawa S, Noda SE, Fujii H, Kono K, Nakano T. Radiotherapy-induced anti-tumor immunity contributes to the therapeutic efficacy of irradiation and can be augmented by CTLA-4 blockade in a mouse model. PLoS One. 2014 Mar 31;9(3):e92572. doi: 10.1371/journal.pone.0092572. eCollection 2014. PMID 24686897
- [Background] Sato H, Suzuki Y, Yoshimoto Y, Noda SE, Murata K, Takakusagi Y, Okazaki A, Sekihara T, Nakano T. An abscopal effect in a case of concomitant treatment of locally and peritoneally recurrent gastric cancer using adoptive T-cell immunotherapy and radiotherapy. Clin Case Rep. 2017 Feb 15;5(4):380-384. doi: 10.1002/ccr3.758. eCollection 2017 Apr. PMID 28396751
- [Background] Kang YK, Boku N, Satoh T, Ryu MH, Chao Y, Kato K, Chung HC, Chen JS, Muro K, Kang WK, Yeh KH, Yoshikawa T, Oh SC, Bai LY, Tamura T, Lee KW, Hamamoto Y, Kim JG, Chin K, Oh DY, Minashi K, Cho JY, Tsuda M, Chen LT. Nivolumab in patients with advanced gastric or gastro-oesophageal junction cancer refractory to, or intolerant of, at least two previous chemotherapy regimens (ONO-4538-12, ATTRACTION-2): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2017 Dec 2;390(10111):2461-2471. doi: 10.1016/S0140-6736(17)31827-5. Epub 2017 Oct 6. PMID 28993052
- [Derived] Mimura K, Ogata T, Nguyen PHD, Roy S, Kared H, Yuan YC, Fehlings M, Yoshimoto Y, Yoshida D, Nakajima S, Sato H, Machida N, Yamada T, Watanabe Y, Tamaki T, Fujikawa H, Inokuchi Y, Hayase S, Hanayama H, Saze Z, Katoh H, Takahashi F, Oshima T, Goel A, Nardin A, Suzuki Y, Kono K. Combination of oligo-fractionated irradiation with nivolumab can induce immune modulation in gastric cancer. J Immunother Cancer. 2024 Jan 30;12(1):e008385. doi: 10.1136/jitc-2023-008385. PMID 38290769

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiotherapy + Nivolumab: Localized short-term radiotherapy (22.5 Gy/5 fractions/5 days, Day 1-5) + nivolumab (starting on Day 15-22, a dose of 3 mg/kg (body weight) or 240 mg/body, every 2 weeks to a total of 6 courses)
  Radiotherapy of 22.5 Gy/5 fractions/5 days was given to a symptomatic lesion or the largest asymptomatic lesion suitable for irradiation from Day 1.
  Nivolumab was administered intravenously starting on Day 15-22 at a dose of 3 mg/kg (body weight) or 240 mg/body every 2 weeks to a total of 6 courses of administration.
Period: Overall Study
Arm/Group | Radiotherapy + Nivolumab
Started | 41
Completed | 22
Not Completed | 19
Not completed — Lack of Efficacy | 16
Not completed — 3 cases did not meet the criteria for nivolumab initiation. | 3

BASELINE CHARACTERISTICS:
Population: A total of 41 patients enrolled in this study were subjected to the safety analysis, and 40 patients, excluding one ineligible patient (72 years old, male), were subjected to the efficacy analysis.
Arm/Group | Radiotherapy + Nivolumab
Number analyzed (Participants) | 41
Age, Continuous [Median (Full Range); unit: years] | 70 [36 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Eligible patients [Count of Participants; unit: Participants] | 40

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate
Description: Analysis item: Disease control rate of non-irradiated target lesions. The rate of patients with a best overall response of stable disease (SD) or better confirmed by 180 days, starting from the start date of radiotherapy. The RECIST Guidelines Version 1.1 was used to determine overall response such as complete response (CR), partial response (PR), SD, and progressive disease (PD) at each imaging time. If imaging is not available, the patient is considered deficient (NE).
Time Frame: 6 months
Population: Since one patient whose target lesions did not meet the selection criteria for this study according to the RECIST guideline version 1.1 was ineligible and was excluded from the efficacy analysis, 40 patients were included in the efficacy analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Radiotherapy + Nivolumab: Single arm study: Localized short-term radiotherapy (22.5 Gy/5 fractions/5 days, Day 1-5) + nivolumab (starting on Day 15-22, a dose of 3 mg/kg (body weight) or 240 mg/body, every 2 weeks to a total of 6 courses).
Arm/Group | Radiotherapy + Nivolumab
Number analyzed (Participants) | 40
Participants | 9

2. Secondary Outcome: Median Survival Time
Description: Overall survival is defined as the period from the start date of radiotherapy until the date of death from any cause or date of last documented survival. In surviving cases, the last date of confirmation of survival is the date of termination. Untraceable cases are terminated on the last date of confirmed survival before the loss of follow-up. At the end of the study period, all enrolled cases are confirmed alive.
Time Frame: From the start date of radiotherapy until the date of death from any cause or date of last documented survival, assessed up to approximately 31 months.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Radiotherapy + Nivolumab
Number analyzed (Participants) | 40
Days | 230 [157 to 330]

3. Secondary Outcome: Safety (Grade and Frequency of Adverse Events)
Description: The frequency of adverse events from all enrolled cases is tabulated by adverse event name and worst grade according to CTCAE ver.4.0. All adverse events are summarized without regard to causal relationships to the study treatment. The frequency and rate of grade 3 or higher adverse events are calculated.
Time Frame: Adverse events were monitored from the start date of radiotherapy until the end of study protocol or death from any cause, and were assessed up to approximately 6 months. All-Cause Mortality was assessed up to approximately 31 months.
Population: The frequency and rate of grade 3 or higher adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiotherapy + Nivolumab
Number analyzed (Participants) | 41
Participants
  Anemia | 8
  Anorexia | 5
  Tumor pain | 3
  Dehydration | 2
  Nausea | 2
  Alkaline phosphatase increased | 1
  Blood bilirubin increased | 1
  Cholecystitis | 1
  Dyspnea | 1
  Febrile neutropenia | 1
  Fever | 1
  Gastric hemorrhage | 1
  Hyperglycemia | 1
  Hyperkalemia | 1
  Hyperuricemia | 1
  Hypoalbuminemia | 1
  Hyponatremia | 1
  Ileus | 1
  Platelet count decreased | 1
  Proteinuria | 1
  Supraventricular tachycardia | 1
  White blood cell decreased | 1
  Lung infection | 1

4. Secondary Outcome: Local Control Rate
Description: Analysis item: Disease control rate of irradiated target lesions. The rate of patients with a best overall response of SD or better confirmed by 180 days, starting from the start date of radiotherapy. The RECIST Guidelines Version 1.1 was used to determine overall response such as CR, PR, SD, and PD at each imaging time. If imaging is not available, the patient is considered NE.
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Radiotherapy + Nivolumab
Number analyzed (Participants) | 40
Participants | 16

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the start date of radiotherapy until the end of study protocol or death from any cause, and were assessed up to approximately 6 months. All-Cause Mortality was assessed up to approximately 31 months.
Arm/Group | Radiotherapy + Nivolumab
All-Cause Mortality (participants affected / at risk) | 28/41
Serious Adverse Events (participants affected / at risk) | 16/41
Other Adverse Events (participants affected / at risk) | 19/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiotherapy + Nivolumab (N=41)
Anemia (Blood and lymphatic system disorders) | 8
Anorexia (Metabolism and nutrition disorders) | 5
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 1
Gastric hemorrhage (Gastrointestinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Platelet count decreased (Investigations) | 1
Proteinuria (Renal and urinary disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
White blood cell decreased (Investigations) | 1
Lung infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Radiotherapy + Nivolumab (N=41)
Fatigue (General disorders) | 9
Aspartate aminotransferase increased (Investigations) | 8
Hypocalcemia (Metabolism and nutrition disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 6
Vomiting (Gastrointestinal disorders) | 6
Alanine aminotransferase increased (Investigations) | 5
Constipation (Gastrointestinal disorders) | 5
Edema limbs (General disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 5
Creatinine increased (Investigations) | 4
Hypertension (Vascular disorders) | 4
Diarrhea (Gastrointestinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/64/NCT03453164/Prot_001.pdf
  • Statistical Analysis Plan (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/64/NCT03453164/SAP_002.pdf
  • Informed Consent Form (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT03453164/ICF_003.pdf